CLINICAL TRIAL: NCT06706180
Title: Motivation for Exercise: A Mood-Based Focus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Michael Otto, Professor Michael Otto, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7628E
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Exercise Motivation
Keywords: Exercise motivation; Exercise for mood
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants do not know that there are two motivational conditions. All outcomes are self-reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise for Mood video (Experimental): The Exercise for Mood intervention is an approximately 11-minute video shown to participants which presents a mood-based motivational frame for exercise and physical activity. Video content focuses on discussions related to the immediate mood benefits from exercise, longer-term cognitive and mental health benefits of exercise, effects of positive affect during exercise, and mood-centered strategies for engaging in regular physical activity, including exercising in diverse locations, exercising with friends, and exercising with music or audiobooks.
  Interventions: Other: Exercise for Mood video
- Exercise for Fitness video (Active Comparator): The Exercise for Fitness intervention is an approximately 11-minute video shown to participants which presents a fitness-based motivational frame for exercise and physical activity. Video content focuses on discussions related to the physical health effects of exercise, including cardiovascular health, increased calorie burning, and overall physical wellbeing. The video also includes recommendations for diversity of exercise, balancing cardiovascular and strength-training activities.
  Interventions: Other: Exercise for Fitness video

INTERVENTIONS:
Other: Exercise for Mood video — As per arm of the same name
  Arms: Exercise for Mood video
Other: Exercise for Fitness video — As per arm of the same name
  Arms: Exercise for Fitness video

SUMMARY:
The goal of this study is to assess the effects of an exercise-related video on exercise motivation and adherence. Specifically, the researchers are studying whether an exercise-for-mood video increase levels of exercise motivation as compared to an exercise-for-fitness video.

DETAILED DESCRIPTION:
This study is designed to evaluate two interventions for exercise motivation: an exercise-for-mood video and an exercise-for-fitness video. After screening to determine eligibility, participants will complete two virtual study appointments, scheduled 10-20 days apart. In Phase 1, participants will first consent to the study and complete the DASS-21, ASI-3, and EMI-2. Participants will then complete an interview-format 7-day Physical Activity Recall (7-day PAR) about their exercise over the past week. Participants are then randomized to either the Fitness or Mood video by the researcher and are assigned to watch the video while on the Zoom meeting, approximately 11 minutes long. After the video, participants complete two short questionnaires about the credibility and usefulness of the video they watched. Finally, participants are briefed on safe exercise habits and given a goal of moderate exercise 4 times per week.

In the Phase 2 appointment, participants complete the EMI-2 and the 7-day PAR about their exercise over the past week. Participants are then debriefed on the intent of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Current PS101 student at Boston University
* A score of 14 or higher on the Perceived Stress Scale (PSS)
* Able to read English to provide informed consent
* Familiarity with a computer keyboard and mouse or a touch screen device
* Access to Zoom video conferencing software

Exclusion Criteria:

* Under age 18
* Known conditions prohibiting exercise adoption as identified by risk scores on the PAR-Q (a score of "yes" on one or more items)
* Presence of anorexia nervosa or atypical anorexia nervosa, or recent (6 month) suicidal ideation
* Score of 13 or lower on the Perceived Stress Scale (PSS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Exercise Motivation | Assessed at Phase 1 appointment and Phase 2 appointment, scheduled 10-20 days apart.
  Exercise Motivations Inventory (EMI-2)

SECONDARY OUTCOMES:
Exercise adherence | Retrospective accounting of the past 7 days, assessed at Phase 1 appointment and Phase 2 appointment, scheduled 10-20 days apart.
  Adherence to an exercise goal of moderate-intensity exercise 4 times per week. Evaluated using the 7-day Physical Activity Recall (7-day PAR).
Mood During Exercise | Assessed at Phase 1 appointment and Phase 2 appointment, scheduled 10-20 days apart
  Mood during most typical, intentional physical activity over the past week, evaluated on the Feeling Scale (FS)
Perceived Exertion during Exercise | Assessed at Phase 1 appointment and Phase 2 appointment, scheduled 10-20 days apart
  Exertion during most typical, intentional physical activity over the past week, evaluated on the Ratings of Perceived Exertion scale (RPE)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of primary aims, de-identified data will be eligible for sharing with investigators requesting such data after completion of a valid data-use agreement.
Supporting Information: Study Protocol
Time Frame: 6 months after publication of the primary outcome.
Access Criteria: Investigators with a valid data-use agreement will be able to access the data.